CLINICAL TRIAL: NCT04363060
Title: Azithromycin With Amoxicillin/Clavulanate Versus Amoxicillin/Clavulanate Alone in COVID-19 Patients With Pneumonia and Hospitalized in a Non-intensive Care Unit Ward (AziA): a Superiority Open-label Randomized Controlled Trial
Brief Title: Azithromycin+Amoxicillin/Clavulanate vs Amoxicillin/Clavulanate in COVID19 Patients With Pneumonia in Non-intensive Unit
Acronym: AziA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC20_0168
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Azithromycin; Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin with amoxicillin/clavulanate (Experimental): Combination of azithromycin during 4 days with amoxicillin/clavulanate during 7 days.
  Interventions: Combination Product: Azithromycin with amoxicillin/clavulanate
- Amoxicillin/clavulanate (Active Comparator): Amoxicillin/clavulanate every day during 7 days.
  Interventions: Drug: amoxicillin/clavulanate

INTERVENTIONS:
Combination Product: Azithromycin with amoxicillin/clavulanate — Patients will receive azithromycin 500 mg on day 1 followed by 250mg per day for the next four days with amoxicillin/clavulanate 1 gr 3 times per day during 7 days. In case of allergy, amoxicillin/clavulanate can be replaced by a third-generation cephalosporin
  Arms: Azithromycin with amoxicillin/clavulanate
Drug: amoxicillin/clavulanate — Patients will receive amoxicillin/clavulanate 1 gr 3 times per day during 7 days. In case of allergy, amoxicillin/clavulanate can be replaced by a third-generation cephalosporin
  Arms: Amoxicillin/clavulanate

SUMMARY:
The global pandemic of novel coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) began in Wuhan, China, in December 2019, and has since spread worldwide.1 As of April 14, 2020, there have been more than 1.5 million reported cases and 124 000 deaths in more than 200 countries. A recent open-label nonrandomized French study reporte that addition of azithromycin to hydroxychloroquine in 6 patients resulted in numerically superior viral clearance (6/6, 100%) compared with hydroxychloroquine monotherapy (8/14, 57%) or control (2/16, 12.5%). Azithromycin alone has never been tested, whereas azithromycin has immunomodulating and anti-inflammatory properties that could theoretically prevent or limit secondary worsening. Our hypothesis is that azithromycin combined with amoxicillin/clavulanate will be superior to amoxicillin/clavulanate alone to obtain viral clearance at Day 6 in COVID-19 patients with pneumonia and hospitalized in a non-intensive care unit ward.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 ans,
* Patient with positive SARS-CoV-2 RT-PCR on nasopharyngeal sample at randomization or within the previous 48 hours,
* Patient with pneumonia diagnosed by thorax CT-scan or echography,
* Patient able to take per os medication,
* Written and signed consent of the patient,
* Patients affiliated with or benefitting from a social security scheme.

Exclusion Criteria:

* Patient hospitalized in intensive care unit,
* Patient who received more than 24 hours of antibiotic treatment for the ongoing episode,
* Chronic renal failure with a Glomerular Filtration Rate < 20ml/min,
* Severe hepatic failure,
* Severe chronic cardiac insufficiency,
* Allergy to macrolides,
* Electrocardiogram showing corrected QT prolongation greater than 470 ms in men and 480 ms in women.
* Life-threatening presentation expected to lead to possible imminent death (based on provider assessment)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of positive SARS-CoV-2 RT-PCR | Day 6
  Rate of positive SARS-CoV-2 RT-PCR on nasopharyngeal sample

SECONDARY OUTCOMES:
Rate of positive SARS-CoV-2 RT-PCR | Day 10
  Rate of positive SARS-CoV-2 RT-PCR on nasopharyngeal sample
Clinical evolution on the World Health Organization Ordinal Scale for Clinical Improvement for COVID-19 | day 6, day 10, and day 30
  Clinical evolution on the WHO Ordinal Scale for Clinical Improvement for COVID-19 score. Scale ranging from 0 to 8 (0:unifected; 8:dead)
Total duration of antibiotic treatment during the 30 days following inclusion | 30 days
  Total duration of antibiotic treatment during the 30 days following inclusion
Number of all-cause mortality during the 30 days following inclusion | 30 days
  Number of all-cause mortality during the 30 days following inclusion
Number of in-hospital mortality during the 30 days following inclusion | 30 days
  Number of in-hospital mortality during the 30 days following inclusion
Number of patients transferred to intensive care unit during the 30-day follow-up | 30 days
  Number of patients transferred to intensive care unit during the 30-day follow-up
Number of days without mechanical ventilation during the 30 days following inclusion | 30 days
  Number of days without mechanical ventilation during the 30 days following inclusion
adverse events attributable to antibiotic treatment during the 30 days following inclusion | 30 days
  adverse events attributable to antibiotic treatment during the 30 days following inclusion
Hospital length of stay during the 30 days following inclusion | 30 days
  Hospital length of stay during the 30 days following inclusion

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Chu Angers, Angers
  - CHD Vendée, La Roche-sur-Yon
  - CHU Poitiers, Poitiers